CLINICAL TRIAL: NCT02210117
Title: A Pilot Randomized Tissue-Based Study Evaluating Anti-PD1 Antibody or Anti-PD1 + Bevacizumab or Anti-PD1 + Anti-CTLA-4 in Patients With Metastatic Renal Cell Carcinoma Who Are Eligible for Cytoreductive Nephrectomy, Metastasectomy or Post-Treatment Biopsy
Brief Title: Nivolumab With or Without Bevacizumab or Ipilimumab Before Surgery in Treating Patients With Metastatic Kidney Cancer That Can Be Removed by Surgery
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0715; NCI-2014-01857 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0715 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-08-04; First posted 2014-08-06 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Kidney Carcinoma; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Ipilimumab; CTLA-4 Antigen; Metastasectomy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (nivolumab, surgery) (Experimental): Patients receive nivolumab IV over 60 minutes on day 1 every 2 weeks for 6 weeks. Approximately 4 weeks later, patients undergo nephrectomy, metastasectomy or biopsy.
  Beginning 4-6 weeks after surgery, patients in all arms who have clinical response, stable disease, or even slight progression of disease to therapy preoperatively, receive maintenance nivolumab IV over 60 minutes on day 1. Cycles repeat every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Other: Laboratory Biomarker Analysis; Procedure: Metastasectomy; Biological: Nivolumab; Procedure: Therapeutic Conventional Surgery
- Arm B (nivolumab, bevacizumab, surgery) (Experimental): Patients receive nivolumab IV over 60 minutes and bevacizumab IV over 90 minutes on day 1 every 2 weeks for 6 weeks. Patients also undergo nephrectomy, metastasectomy or biopsy as in Arm A.
  Beginning 4-6 weeks after surgery, patients in all arms who have clinical response, stable disease, or even slight progression of disease to therapy preoperatively, receive maintenance nivolumab IV over 60 minutes on day 1. Cycles repeat every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy; Other: Laboratory Biomarker Analysis; Procedure: Metastasectomy; Biological: Nivolumab; Procedure: Therapeutic Conventional Surgery
- Arm C (nivolumab, ipilimumab, surgery) (Experimental): Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes on day 1 every 3 weeks for 6 weeks. Patients also undergo nephrectomy, metastasectomy or biopsy as in Arm A.
  Beginning 4-6 weeks after surgery, patients in all arms who have clinical response, stable disease, or even slight progression of disease to therapy preoperatively, receive maintenance nivolumab IV over 60 minutes on day 1. Cycles repeat every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biopsy; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Procedure: Metastasectomy; Biological: Nivolumab; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm B (nivolumab, bevacizumab, surgery)
Procedure: Biopsy — Undergo biopsy
  Other Names: Bx
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm C (nivolumab, ipilimumab, surgery)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Metastasectomy — Undergo metastasectomy
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Procedure: Therapeutic Conventional Surgery — Undergo nephrectomy

SUMMARY:
This randomized pilot early phase I trial studies the side effects and how well nivolumab alone works compared to nivolumab with bevacizumab or ipilimumab before surgery in treating patients with kidney cancer, also referred to as renal cell cancer, that has spread to another place in body and can be removed by surgery. Immunotherapy with monoclonal antibodies, such as nivolumab, bevacizumab, and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Safety and tolerability of therapy with nivolumab or nivolumab + bevacizumab or nivolumab + ipilimumab in metastatic renal cell carcinoma (mRCC) in the context of presurgical or prebiopsy therapy.

SECONDARY OBJECTIVES:

I. To study immunological changes in tumor tissues and peripheral blood in response to nivolumab versus (vs.) nivolumab + bevacizumab vs nivolumab + ipilimumab in renal cell carcinoma (RCC) therapy.

II. To assess the efficacy of presurgical nivolumab or nivolumab + bevacizumab or nivolumab + ipilimumab therapy in RCC by evaluating objective response rate, duration of response, and progression free survival, and overall survival.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Patients receive nivolumab intravenously (IV) over 60 minutes on day 1 every 2 weeks for 6 weeks. Approximately 4 weeks later, patients undergo nephrectomy, metastasectomy or biopsy.

ARM B: Patients receive nivolumab IV over 60 minutes and bevacizumab IV over 90 minutes on day 1 every 2 weeks for 6 weeks. Patients also undergo nephrectomy, metastasectomy or biopsy as in Arm A.

ARM C: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes on day 1 every 3 weeks for 6 weeks. Patients also undergo nephrectomy, metastasectomy or biopsy as in Arm A.

Beginning 4-6 weeks after surgery, patients in all arms who have clinical response, stable disease, or even slight progression of disease to therapy preoperatively, receive maintenance nivolumab IV over 60 minutes on day 1. Cycles repeat every 4 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and 86 days, every 3 months for 2 years, every 6 months for 1 year, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must give written informed consent prior to initiation of therapy, in keeping with the policies of the institution; patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of the study and the risks associated with the therapy
* Patients with histologically or cytologically confirmed metastatic clear cell RCC who are eligible for cytoreductive nephrectomy, metastasectomy or post-treatment biopsy; diagnosis must be confirmed by pathologist review of screening biopsy; the determination of resectability will ultimately lie in the clinical judgment of the urologist and medical oncologist involved in the care of the patient
* Patients must have measurable disease and is defined as a lesion that can be accurately measured on the long axis with a minimum size of 10 mm or a lymph node that can be accurately measured along the short axis of a minimum size of 15 mm (computed tomography [CT] scan slice thickness can be no greater than 5 mm)
* Patients can have had prior treatment for RCC including prior surgery, radiation therapy, immunotherapy with interleukin (IL)-2 or interferon (but not anti-programmed cell death [PD]1 or anti-cytotoxic T-lymphocyte-associated protein 4 [CTLA-4]), target therapy with receptor tyrosine kinase (RTK) inhibitors/mammalian target of rapamycin (mTOR) inhibitors, such as sunitinib, sorafenib, pazopanib, axitinib, everolimus, and temsirolimus (but not bevacizumab) or chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Absolute neutrophil count >= 1,500/uL within 14 days of the first dose of study drug
* Platelets >= 100,000/uL within 14 days of the first dose of study drug
* Hemoglobin (Hgb) > 9.0 g/dL (may be transfused or receive epoetin alfa [e.g., Epogen] to maintain or exceed this level) within 14 days of the first dose of study drug
* Total bilirubin =< 1.5 mg/dl within 14 days of the first dose of study drug
* Serum creatinine =< 1.5 times the upper limit of normal or estimated creatinine clearance (CrCl) > 40 mL/min within 14 days of the first dose of study drug
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and/or alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal for patients without evidence of liver metastases, AST (SGOT) and/or ALT (SGPT) =< 5 x institutional upper limit of normal for patients with documented liver metastases within 14 days of the first dose of study drug
* Mild autoimmune conditions (such as localized psoriasis) requiring minimal treatment or systemic autoimmune conditions well controlled by target agents such as an anti-IL-17 that do not affect overall immune system
* Patients with a history of Hashimoto's thyroiditis only requiring hormone replacement, type I diabetes, or conditions not expected to recur in the absence of an external trigger are allowed to participate
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug
* Women must not be breastfeeding
* WOCBP must agree to follow instructions for method(s) of contraception from the time of enrollment for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 30 days (duration of ovulatory cycle) for a total of 23 weeks post treatment completion
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug (s) plus 5 half-lives of study drug (s) plus 90 days duration of sperm turnover for a total of 31 weeks post-treatment completion
* Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements; however WOCBP must still undergo pregnancy testing as described; investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy; investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception; highly effective methods of contraception have a failure rate of < 1% per year when used consistently and correctly; at a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below: HIGHLY EFFECTIVE METHODS OF CONTRACEPTION:

  * Male condoms with spermicide
  * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partner
  * Nonhormonal IUDs, such as ParaGard
  * Tubal ligation
  * Vasectomy
  * Complete abstinence

    * Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs; abstinence is only acceptable when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, profession of abstinence for entry into a clinical trial, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests; acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence; LESS EFFECTIVE METHODS OF CONTRACEPTION:

  * Diaphragm with spermicide
  * Cervical cap with spermicide
  * Vaginal sponge
  * Male condom without spermicide

    * A male and female condom must not be used together
  * Progestin only pills by WOCBP subject or male subject's WOCBP partner
  * Female condom

    * A male and female condom must not be used together

Exclusion Criteria:

* Any other malignancy from which the patient has been disease-free for less than 2 years, except for non-melanoma skin cancer, in situ carcinoma of any site
* Patients who have organ allografts
* Patients who have had a major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to first dose of study drug; or anticipation of need for major surgical procedure during the course of the study (other than defined by protocol); or fine needle aspirations or core biopsies within 7 days prior to first dose of study drug
* Known or suspected autoimmune disease; patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]) are excluded from this study; any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug; inhaled steroids and adrenal replacement steroids doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS); positive test for hepatitis B virus (HBV) using HBV surface antigen (HBV sAg) test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection
* Any underlying medical condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea
* Patients who have had a history of acute diverticulitis, abdominal fistula, gastrointestinal perforation, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation, should be excluded from the study
* Patients who have a primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, history of stroke within the past year
* History of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of > 140/90 mmHg) at the time of enrollment, New York Heart Association (NYHA) grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease or symptomatic peripheral vascular disease
* Patients who have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Patients who have proteinuria at baseline; patients who are unexpectedly discovered to have >= grade 2 proteinuria at baseline routine urinalysis should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate =< 1 g of protein/24 hour (hr) to allow participation in the study
* Patients who have uncontrolled hypertension (systolic > 140 mmHg and/or diastolic > 90 mmHg); it is permissible to start treatment for hypertension prior to randomization
* Patients who are on high dose steroid (e.g. > 10 mg prednisone daily or equivalent) or other more potent immune suppression medications (e.g. infliximab)
* Patients who have had flu, hepatitis, or other vaccines within a month prior to initiation of study drugs
* Patients who have clinical history of coagulopathy, bleeding diathesis or thrombosis within the past year
* Patients who have serious, non-healing wound, ulcer, or bone fracture
* Pregnancy (positive pregnancy test) or lactation
* Patients must not have received prior anticancer therapy with bevacizumab, anti-CLTA-4, or anti-PD1 for renal cell carcinoma; patients receiving any concomitant systemic therapy for renal cell cancer are excluded
* Patients must not be scheduled to receive another experimental drug while on this study
* Patients who require ongoing anticoagulation will be excluded; only aspirin will be permitted; pre and post-surgical prophylactic anti-coagulation treatment is permitted
* Patients must not require total parenteral nutrition with lipids
* Any patients who cannot be compliant with the appointments required in this protocol must not be enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events, defined any grade 3 or higher adverse event that is possibly, probably, or definitely related to any therapy received on this protocol | 6 weeks
  Descriptive statistical analyses will be performed to summarize the overall toxicity rate and individual adverse event rates including summary tables, scatter-plots, box-plots, proportions, median, means, and standard deviations.

SECONDARY OUTCOMES:
Immunological changes in tumor tissues and peripheral blood | Baseline to up to week 4
  Descriptive statistical analyses will be performed to summarize the immunological changes, including summary tables, scatter-plots, box-plots, proportions, median, means, and standard deviations. A mixed model accounting for patient effects will be used to analyze the longitudinal data on immunological values over time.
Objective response rates | Up to 5 years
  Descriptive statistical analyses will be performed to summarize the response rates including summary tables, scatter-plots, box-plots, proportions, median, means, and standard deviations.
Duration of response | Up to 5 years
  Will be estimated with the methods of Kaplan and Meier.
Progression-free survival | Up to 5 years
  Progression-free survival will be estimated with the methods of Kaplan and Meier.
Overall survival | Up to 5 years
  Will be estimated with the methods of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Padmanee Sharma, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org